CLINICAL TRIAL: NCT03746743
Title: Severity Index of Neonatal Septicemia of Cases Admitted at Neonatal Intensive Care Units at CHILDREN'S HOSPITAL, CAIRO UNIVERSITY and at ELGALAA Children's MILITARY HOSPITAL Using Score for Neonatal Acute Physiology (SNAP) II
Brief Title: Severity Index of Neonatal Septicemia Using Score for Neonatal Acute Physiology (SNAP) II
Acronym: SNAP
Status: Completed | Type: Observational
Sponsor: Ahmed Mahmoud Ali Ali Youssef (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mahmoud Ali Ali Youssef, Doctor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: SNAP II Score
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Neonatal SEPSIS
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm neonates: Neonates born between 32 and 37 weeks gestation
  Interventions: Diagnostic Test: score for neonatal sepsis
- Fullterm neonates: Neonates born at or after 37 weeks gestation
  Interventions: Diagnostic Test: score for neonatal sepsis

INTERVENTIONS:
Diagnostic Test: score for neonatal sepsis — score for neonatal sepsis to predict morbidity

SUMMARY:
To determine the effect of Score for Neonatal Acute Physiology II as a Predictor of Mortality and Organ Dysfunction in Neonates with Septicemia in the Neonatal Intensive Care Units at CHILDREN'S HOSPITAL, CAIRO UNIVERSITY and at ELGALAA Children's MILITARY HOSPITAL.

DETAILED DESCRIPTION:
This study will be conducted at the Neonatal intensive care Units at CHILDREN'S HOSPITAL, CAIRO UNIVERSITY and at ELGALAA Children's MILITARY HOSPITAL.

Population of study & disease condition:

Neonates with septicemia admitted to NICUs in CHILDREN'S HOSPITAL, CAIRO UNIVERSITY and in ELGALAA Children's MILITARY HOSPITAL.

Inclusion criteria:

1. Type of patient: Neonates with septicemia.
2. Age of patient: From 0-28 Days.
3. Sex: males and females.

Exclusion criteria:

1. Neonates with proved inborn error of metabolism.
2. Neonates with multiple congenital anomalies.
3. Neonates with severe birth asphyxia (APGAR score <4 at 5 minutes).

Methodology in details:

We will have 2 groups, each of them 50 neonates with septicemia. One group of premature neonates (32-36 weeks), the other group of full term neonates (>37 weeks).

All included Patients will be subjected to the following:

1. Full history with emphasis of relevant data as follows:

   Date of birth, gestational age (AGA or SGA), gender, day of sepsis onset.
2. Clinical assessment:

   Full systems examination.
3. Diagnosis of sepsis:

   * By abnormal Total leucocytic count or I/T ratio or CRP with clinical Suggestion (poor feeding, hepatomegaly, apnea, tachypnea, lethargy, …).
   * Confirm diagnosis by blood culture.

   Sepsis will be considered severe if the neonate has sepsis plus one of the following: 1) cardiovascular organ dysfunction (hypotension or need for vasoactive drug) 2) 2 of the following (metabolic acidosis, increase lactic acid, oliguria, Prolonged capillary refill time) 3) Organ dysfunction (respiratory, renal, neurologic, hematologic).
4. SNAP II score:

   For all neonates included in the study and its data collection within 24 hours from onset of sepsis, in the form of:
   * Lowest mean blood pressure.
   * Worst ratio of pao2/fio2
   * Lowest temperature.
   * Lowest serum PH.
   * Occurrence of multiple seizures.
   * Urine output<1 ml/kg/hour.
5. Follow up:

   Follow up all neonates included in the study for 14 days: for morbidity and mortality.
6. Diagnosis of organ dysfunction:

Respiratory: by CXR and clinical examination. CVS: by blood pressure, capillary refill time, shock and need for inotropes. Renal: by urine output, kidney function tests. Hematology: by picture of DIC or pancytopenia. Neurology: by seizures, dilated fixed pupil.

Possible Risk:

None.

Primary outcomes:

Using Score for Neonatal Acute Physiology II as a Predictor of Mortality and Organ Dysfunction in Neonates with Septicemia.

Secondary outcomes:

Early anticipation of clinical manifestations of sepsis which will correlate most with poor outcome.

Sample size:

100 Neonates with septicemia admitted to NICUs in CHILDREN'S HOSPITAL, CAIRO UNIVERSITY and in ELGALAA Children's MILITARY HOSPITAL.

ELIGIBILITY:
Inclusion Criteria:

1. Type of patient: Neonates with septicemia.
2. Age of patient: From 0-28 Days.
3. Sex: males and females.

Exclusion Criteria:

1. Neonates with proved inborn error of metabolism.
2. Neonates with multiple congenital anomalies.
3. Neonates with severe birth asphyxia (APGAR score <4 at 5 minutes).

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with septicemia admitted to NICUs in CHILDREN'S HOSPITAL, CAIRO UNIVERSITY and in ELGALAA Children's MILITARY HOSPITAL.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Using Score for Neonatal Acute Physiology II as a Predictor of Mortality and Organ Dysfunction in Neonates with Septicemia. | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Early anticipation of clinical manifestations of sepsis which will correlate most with poor outcome. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nermin R Mohamed, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty Of medicine Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No